CLINICAL TRIAL: NCT06648941
Title: Evaluation of Medial Supraspinatus Muscle Release in Treatment of Retracted Rotator Cuff Tear
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Hemaid Mostafa, Mustafa hemaid, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-08-01MD; no one (Other: no one)
Record Dates: First submitted 2024-10-01; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Rotator Cuff Tears of the Shoulder
Keywords: rotator cuff tear; supraspinatus muscle
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Myotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supraspinatus muscle release (Other): supraspinatus muscle release in retracted rotator cuff tear
  Interventions: Procedure: Muscle release

INTERVENTIONS:
Procedure: Muscle release — supraspinatus muscle release

SUMMARY:
- Introduction Rotator cuff tears are a prevalent cause of shoulder pain and dysfunction, particularly among individuals engaged in repetitive overhead activities or advancing in age. The supraspinatus muscle, integral to shoulder function, initiates abduction and provides essential stability to the glenohumeral joint. When the supraspinatus tendon tears and retracts, surgical intervention is often necessary to restore function and alleviate symptoms. (1) Traditional surgical approaches for retracted rotator cuff tears typically involve reattaching the tendon to the greater tuberosity of the humerus. However, severe retraction can lead to challenges during repair, including increased tension on the repair site, potentially compromising healing and increasing the risk of re-tears. • Partial Repair with or without Augmentation: In cases of moderate retraction where complete tendon mobilization is challenging, a partial repair combined with augmentation techniques (e.g., patch augmentation, autografts, allografts) may be considered to optimize tendon-to-bone healing.

• Tendon Transfer: For massive irreparable tears or poor tendon quality, tendon transfer procedures (e.g., transferring the teres minor or lower trapezius tendon) may be necessary to restore function and shoulder stability. (2) To address these challenges, medial release of the supraspinatus tendon from its attachment on the medial border of the scapula has emerged as a promising technique.

Medial release involves detaching the supraspinatus tendon from its scapular attachment and mobilizing it medially. This technique aims to reduce tension at the repair site, allowing for better tendon apposition and potentially improving healing outcomes. Proponents suggest that medial release enhances biomechanical strength and reduces the risk of postoperative complications such as re-tears. However, the technique's optimal application, outcomes, and comparative effectiveness against traditional repair methods remain subjects of ongoing research and debate within the orthopedic community. (3)

Given the complexity and variability of retracted rotator cuff tears, a systematic evaluation of medial release is crucial to clarify its efficacy, safety, and role in surgical management. This protocol outlines a comprehensive framework for evaluating medial release of the supraspinatus tendon in the repair of retracted rotator cuff tears. The study aims to provide evidence-based insights that can guide surgical decision-making, improve patient outcomes, and advance the field of shoulder surgery.

Furthermore, medial release may enhance the biomechanical integrity of the repair. By optimizing tendon positioning and tension during repair, it could improve the mechanical strength of the repair construct. This aspect is crucial for achieving durable outcomes and preventing repair failure over time..

ELIGIBILITY:
Inclusion Criteria

* Adults aged 35-65 years
* Diagnosed with retracted rotator cuff tear confirmed by MRI
* Failed conservative treatment for at least 6 months
* Informed consent provided

  - Exclusion Criteria
* Previous fracture around shoulder on the affected side
* shoulder infection on the affected side
* Axillary nerve injury
* Previous shoulder surgery on the affected side

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in pain score ( vas) score | one year
  Improvement in pain score ( vas) score at 12 months.

OTHER OUTCOMES:
Rate of re-tear | one year
Incidence of complications (infection, stiffness) | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt sohag, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Evaluation of medial supraspinatus muscle release in retracted rotator cuff tear
Supporting Information: CSR
Time Frame: one year

REFERENCES:
- [Background] Burkhart SS, Danaceau SM, Pearce CE Jr. Arthroscopic rotator cuff repair: Analysis of results by tear size and by repair technique-margin convergence versus direct tendon-to-bone repair. Arthroscopy. 2001 Nov-Dec;17(9):905-12. doi: 10.1053/jars.2001.26821. PMID 11694920
- [Background] Gerber C, Fuchs B, Hodler J. The results of repair of massive tears of the rotator cuff. J Bone Joint Surg Am. 2000 Apr;82(4):505-15. doi: 10.2106/00004623-200004000-00006. PMID 10761941
- [Background] Boileau P, Brassart N, Watkinson DJ, Carles M, Hatzidakis AM, Krishnan SG. Arthroscopic repair of full-thickness tears of the supraspinatus: does the tendon really heal? J Bone Joint Surg Am. 2005 Jun;87(6):1229-40. doi: 10.2106/JBJS.D.02035. PMID 15930531